CLINICAL TRIAL: NCT02785731
Title: ANG-001 Pelvic Mass Training Study: Evaluation of Multiple Circulating Tumor Cell-derived RNA Markers to Estimate Risk of Ovarian Cancer in Patients Presenting With a Pelvic Mass.
Brief Title: Evaluation of Multiple Biomarkers to Estimate Risk of Ovarian Cancer in Patients With a Pelvic Mass.
Status: Completed | Type: Observational
Sponsor: Angle plc (Industry)
Collaborators: Medical University of Vienna (Other); Charite University, Berlin, Germany (Other); Vivantes Netzwerk für Gesundheit GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: ANG-001
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Ovarian Neoplasms
Keywords: pelvic mass; ovarian cancer; gynecological cancer; risk prediction
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection; Phlebotomy; Laparotomy; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All excess components (i.e. serum, plasma, RNA, DNA, cells, etc.) generated from the peripheral blood samples collected for research testing under this study be stored frozen at the Medical University of Vienna for up to 10 years for possible use in future research, including but not limited to, serum biomarker analyses, genomic evaluations and genetic studies pertaining to cancer and other disease processes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with a pelvic mass: Women diagnosed with a pelvic mass (defined as a simple, complex or a solid ovarian cyst / pelvic mass) who are scheduled for a laparotomy or laparoscopy for removal of the pelvic mass. Must have a pelvic imaging study performed within 60 days prior to surgery and a research blood draw within 60 days prior to surgery.
  Interventions: Procedure: Pelvic imaging; Procedure: Blood draw; Procedure: laparotomy or laparoscopy

INTERVENTIONS:
Procedure: Pelvic imaging — Within 60 days prior to the pelvic mass evaluation procedure, each subject must have a pelvic imaging study (e.g. ultrasound, CT scan, MRI, etc.) conducted and read to visualize the pelvic mass according to the current standard of care. Results of the pelvic imaging study(ies) will be recorded.
  Other Names: pelvic ultrasound; CT scan; MRI scan
Procedure: Blood draw — Within 60 days prior to, or on the day of the pelvic mass surgery, collect up to 35mL of whole blood into one 5mL SST tube, which must be drawn first, followed by three separate 10mL EDTA tubes.
  Other Names: phlebotomy
Procedure: laparotomy or laparoscopy — A laparotomy or laparoscopic procedure will be performed by a qualified individual for excision of the pelvic mass. Representative tissue samples will be taken from the excised pelvic mass and evaluated in pathology departments within each institution according to institutional guidelines. Results from the histopathological evaluation will be recorded, including the final diagnosis along with histological sub-type, and if available, stage and grade of cancer where disease is identified.

SUMMARY:
ANGLE has developed the Parsortix™ Cell Separation System (Parsortix), an automated system capable of harvesting rare circulating cells for analysis from a sample of peripheral blood based on cellular size and deformability. In a small pilot study, scientists at the Medical University of Vienna demonstrated that measurement of a combination of mRNA markers extracted from CTCs captured using the Parsortix system could be used to identify women with ovarian cancer. This study is designed to provide specimens for optimization of an assay using clinical and biomarker information (i.e. demographics, imaging results and/or serum tumor markers) in combination with mRNA extracted from rare cells in the blood of women presenting with a pelvic mass for the detection of malignancy.

Primary Objective: Optimization of an assay for the differentiation of women with benign pelvic masses from those with malignant pelvic masses using mRNA markers extracted from CTCs isolated from whole blood. Multiple serum tumor markers and mRNA markers will be measured, and the results will be compared to the actual clinical diagnosis made for each patient through other recognized methods (e.g. histopathology). The blood samples collected in the course of this study will be used to finalize the selection of mRNA and/or serum tumor markers to be evaluated in future prospective studies.

Exploratory Objective: Use statistical modeling to determine the need for and/or preliminary design of a mathematical algorithm to combine the multiple serum tumor and/or mRNA markers for estimation of the risk of ovarian cancer.

DETAILED DESCRIPTION:
This study is exploratory in nature and is designed to be hypothesis generating to support the design of future studies. A total of 200 women diagnosed with a pelvic mass (defined as a simple, complex or a solid ovarian cyst / pelvic mass) who are scheduled for a laparotomy or laparoscopy for removal of the pelvic mass will be enrolled for evaluation of the primary and exploratory endpoints. An initial evaluation of the data will be conducted after identification of 15 evaluable subjects with histopathologically confirmed ovarian cancer. It is estimated that 50 - 100 subjects will be required to obtain a minimum of 15 evaluable subjects with histopathologically confirmed ovarian cancer. The remainder of the women enrolled (expected to be ~100 - 150 subjects) will be used to verify the findings from the initial evaluation (i.e. correlation of the markers with the absence or presence of malignancy) and to refine the assay/algorithm.

Within 60 days prior to surgery, each subject must have a pelvic imaging study (e.g. ultrasound, CT scan, MRI, etc.) conducted and read to visualize the pelvic mass according to the current standard of care. Results of the pelvic imaging study(ies) will be recorded.

Within 60 days prior to, or on the day of the pelvic mass surgery, collect up to 35mL of peripheral blood into one 5mL SST tube, which must be drawn first, followed by three separate 10mL EDTA tubes. Serum from SST tube will be prepared at the local study center and used for protein biomarker testing. The EDTA tubes will be shipped to the Medical University of Vienna, where the blood will be pooled and equal volumes processed using two different separation methods on the Parsortix™ system to capture and harvest rare cells. The harvested material from the EDTA tubes will be lysed, and total RNA will be extracted from the cell lysate for evaluation of multiple gene targets using quantitative PCR (qPCR).

Laparotomy or laparoscopy for removal of the pelvic mass will be performed by a qualified individual. Tissue samples will be sent to the local pathology department for histological examination in accordance with standard institutional practices. Results of the histopathological evaluation will be recorded, including the final diagnosis along with histological sub-type, and if available, stage and grade of ovarian cancer where disease is identified.

Subjects will be considered negative for ovarian cancer:

* if the subject undergoes surgery and no mass is identified, or;
* if the histopathological findings are negative for cancer (i.e. benign conditions).

Subjects will be considered positive for ovarian cancer:

* if the histological examination of the tissue taken at the time of surgery confirms the presence of ovarian, primary peritoneal and/or fallopian tube cancers.

For the purposes of enrollment, subjects diagnosed with a malignancy other than an ovarian cancer as well as those diagnosed with low malignant potential (LMP) / borderline tumors will not be counted as an ovarian cancer. However, two separate analyses of the final study data will be conducted: one where subjects diagnosed with other cancers are excluded from the analysis of the primary endpoint and the subjects diagnosed with LMP / borderline tumors are classified as being negative for malignancy, and a second where subjects diagnosed with other cancers and those diagnosed with LMP / borderline tumors are classified as being positive for malignancy.

Demographical and clinical data may be summarized using descriptive statistics. Continuous variables may be summarized using the number of observations, mean, standard deviation, coefficient of variation, median, and range as appropriate. Categorical values may be summarized using the number of observations and percentages as appropriate.

The association of the markers (i.e. serum protein markers and mRNA markers) with the histopathological diagnosis will be assessed using appropriate statistical methods (e.g., logistic regression, analysis of variance [ANOVA], etc.), depending on the endpoints. Analyses may be performed within and between various histopathological diagnosis sub-groups. Other clinical covariates (such as imaging results and subject demographics) may also be included in the modeling.

An initial evaluation of the correlation of the markers with the histopathological diagnosis will be performed after the identification of 15 subjects with histopathologically verified ovarian cancer. The final cohort of patients will be used to verify the findings from the initial evaluation (i.e. correlation of the markers with the absence or presence of malignancy) and to refine the assay/algorithm. Bootstrap analyses may be utilized on the entire set of 200 subjects to finalize an assay/algorithm for further study.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age;
* Documented evidence of a pelvic mass by imaging;
* Selected to undergo laparotomy or laparoscopy based on the finding of a pelvic mass (defined as a simple, complex or a solid ovarian cyst / pelvic mass);
* Willing and able to provide written informed consent prior to the blood collection.
* Suitable venous access and healthy enough (as determined by the treating physician) to provide required whole blood sample.

Exclusion Criteria:

* Known pregnancy;
* Subjects receiving cytotoxic chemotherapies;
* Previous malignancy within the past 5 years, excluding skin cancers (squamous cell or basal cell);
* Unwilling or unable to follow protocol requirements or to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with a pelvic mass (defined as a simple, complex or a solid ovarian cyst / pelvic mass) who are scheduled for a laparotomy or laparoscopy for removal of the pelvic mass.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Histopathological diagnosis | Within 30 days after biopsy or surgical procedure to evaluate pelvic mass
  Tissue samples taken from the pelvic mass will be evaluated in the local institutional pathology department according to institutional guidelines. Results from the histopathological evaluation, including the final diagnosis (i.e. benign, malignant, etc.), histopathology description, and, if malignant, clinical or surgical staging and tumor subtype, will be recorded.
Presence or absence of circulating tumor cells | Up to 60 days prior to surgical procedure to evaluate pelvic mass
  Blood from EDTA tubes will be pooled and processed on the Parsortix System to capture and harvest rare cells. The captured rare cells will be eluted (harvested) and lysed, and total RNA will be extracted from the cell lysate for evaluation of multiple gene targets using quantitative PCR (qPCR).
Serum protein markers | Up to 60 days prior to surgical procedure to evaluate pelvic mass
  Serum from SST tube will be used for protein biomarker testing.

CONTACTS AND LOCATIONS:
Overall Officials: Shane Booth, Ph.D., Study Director — Angle plc
Locations (5):
- Medical University of Vienna, Vienna, Austria
- Germany (4):
  - Vivantes Auguste-Viktoria-Klinikum, Berlin
  - Vivantes-Klinikum Neukölln, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Vivantes Humboldt-Klinikum, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obermayr E, Castillo-Tong DC, Pils D, Speiser P, Braicu I, Van Gorp T, Mahner S, Sehouli J, Vergote I, Zeillinger R. Molecular characterization of circulating tumor cells in patients with ovarian cancer improves their prognostic significance -- a study of the OVCAD consortium. Gynecol Oncol. 2013 Jan;128(1):15-21. doi: 10.1016/j.ygyno.2012.09.021. Epub 2012 Sep 24. PMID 23017820
- [Background] Obermayr E, Sanchez-Cabo F, Tea MK, Singer CF, Krainer M, Fischer MB, Sehouli J, Reinthaller A, Horvat R, Heinze G, Tong D, Zeillinger R. Assessment of a six gene panel for the molecular detection of circulating tumor cells in the blood of female cancer patients. BMC Cancer. 2010 Dec 3;10:666. doi: 10.1186/1471-2407-10-666. PMID 21129172
- See also: Study Sponsor Website — http://www.angleplc.com
- See also: Charite Comprehensive Cancer Center Website — http://cccc.charite.de/en/
- See also: Medical University of Vienna Website — http://www.meduniwien.ac.at/homepage/1/homepage/